CLINICAL TRIAL: NCT00350064
Title: Impact of Exercise Training Intensity on Abdominal Visceral Fat and Risk Factors Associated With the Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Arthur Weltman/Principal Investigator, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UVAHIC11145
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Obesity; Exercise; Diabetes; Physical Activity
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Motor Activity; Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise Training — 16 weeks of aerobic exercise training at two different intensities

SUMMARY:
The purpose of this study is to determine if sixteen weeks of high intensity physical training is more effective than sixteen weeks of low intensity physical training in reducing abdominal fat and lowering risk factors associated with the metabolic syndrome. Another aim of this study is to determine if high intensity physical training improves cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have meet the definition of the metabolic syndrome (based on IDF consensus statement).
* Screening biochemical tests of liver, kidney, hematologic, metabolic (below) and thyroid function must be normal.
* The volunteer must be willing to:

  1. visit the outpatient GCRC or clinic once monthly for 16 weeks of intervention,
  2. participate in supervised exercise training (if assigned) and
  3. enter the inpatient GCRC for 2-3 days of more intensive studies at baseline and after 16 weeks of intervention. The subject must provide voluntary and fully informed written consent.

Exclusion Criteria:

* Type 1 diabetes,
* drug or alcohol abuse,
* psychosis,
* severe or untreated depression,
* dementia, polycythemia (hematocrit > 55%),
* clinically symptomatic coronary artery,
* pulmonary or orthopedic disease (which would disallow exercise training),
* history of vascular or peripheral nerve trauma,
* lymph node dissection,
* anemia, uncontrolled hypertension (> 160/105 untreated or > 145/95 treated),
* allergic to octafluoropropane, or nitroglycerine,
* weight loss or gain of 2 kg or more within the preceding 10 days,
* investigational drug use within five biological half-lives,
* treatment with ACE inhibitors or ARBs, thiazolindiones,
* 1st or 2nd generation anti-psychotics insulin, or Viagra,
* unwillingness to provide written informed voluntary consent,
* pregnant, breast feeding or use hormonal birth control.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2004-04; Primary Completion 2006-06 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Change in Abdominal Visceral Fat | before and after 16 weeks

SECONDARY OUTCOMES:
VO2peak | before and after 16 weeks
% Body Fat | before and after 16 weeks
Insulin | before and after 16 weeks
FFA | before and after 16 weeks
Glucose | before and after 16 weeks
Hba1c | before and after 16 weeks
Cholesterol | before and after 16 weeks
CRP | before and after 16 weeks
IL6 | before and after 16 weeks
TNF | before and after 16 weeks
Homocysteine | before and after 16 weeks
Adiponectin | before and after 16 weeks
Adhesion Molecules | before and after 16 weeks
Endothelial Function | before and after 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Weltman, PhD, Principal Investigator — University of Virginia; Brian A Irving, PhD, Study Director — University of Virginia
Locations (1):
- University of Virginia General Clinical Research Center, Charlottesville, Virginia, United States